CLINICAL TRIAL: NCT04083248
Title: Building Self-regulation Capacity in AA T2DM Women: Feasibility of an Ecological Momentary Intervention
Brief Title: Building Self-regulation Capacity in AA T2DM Women: Feasibility of EMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Risks to subjects due to COVID-19
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Chicago (Other)
Responsible Party: Principal Investigator, Cynthia Fritschi, PhD, Associate Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-0922; P30DK092949 (NIH)
Record Dates: First submitted 2019-08-30; First posted 2019-09-10 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes; Self-regulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility group (Experimental): Intervention components:
  Personalized group diabetes education.
  Fitbit Charge 3 wrist activity monitor for real-time monitoring of steps, active minutes and heart rate. The Fitbit will be used by the women to set activity goals, self-assess their progress and aid in motivation to be more active.
  Freestyle Libre (Abbott Labs, Alameda, CA) Personal CGM (FDA approved). The Libre CGM will be used to self-monitor glucose goals and monitor the real-time effects of activity and eating choices by the women.
  Final guided interview for study acceptability and feasibility. The interviews will be audiotaped, transcribed. Thematic content analyses will be performed.
  Interventions: Behavioral: Feasibility group

INTERVENTIONS:
Behavioral: Feasibility group — Same as arm description

SUMMARY:
In African-Americans, the incidence of type 2 diabetes (T2DM) is ~14%. Adherence to crucial diabetes self-management (DSM) behaviors, such as engaging in physical activity (PA) is dangerously low among AA women living in disadvantaged neighborhoods. These women manage numerous chronic challenges (daily discrimination, poverty, and violence), which drain the internal energy needed for DSM. The ability to self-regulate (modify one's behaviors based on the requirements of a situation) has been associated with adherence to health behaviors, including diet and PA. This 6-week ecological momentary intervention (EMI) feasibility study has been developed to reduce energy needs of DSM through use of self-regulation strategies delivered in real-time, in the real-world setting. Twenty-six AA women will receive personalized diabetes education over two days. They will be given a personalized activity prescription and a Fitbit wrist activity monitor. During the following two weeks, they will get a personal continuous glucose monitor (CGM) and individualized "cue cards" for simple behaviors they can try when glucose levels are too high. The intervention is grounded in self-regulation theory, and targets core self-regulation components, including self-monitoring/assessment, mental contrasting of target values with actual values, and goal-setting/review. The aim for this application is to Determine the feasibility and acceptability of an ecological momentary intervention, consisting of continuous glucose monitoring, activity tracking, and personalized cue cards with behavioral choices (eating/activity) driven by the results of glucose levels. Impact: Real-time feedback on the effects of activity and eating behaviors will enable patients to make choices and see results immediately. Our intervention will offer low-income African-American women opportunities to enact behaviors in their momentary environment, and will encourage autonomous motivation for PA uptake, and improving blood glucose control. Findings from this study will have an important positive impact on our ability to create tailored, EMIs among low-income adults who have limited access to diabetes specialty care and education.

DETAILED DESCRIPTION:
All visits will take place at the University of Illinois at Chicago (UIC) College of Nursing Clinical Diabetes and Exercise Laboratory. At time 1 (T1), participants will complete baseline assessments. Participants will complete health and biological assessments, including measures of glucose control (A1C), body mass index (BMI) and a diabetes health history, including, diabetes knowledge, and current DSM behaviors. The investigators will collect assessments of autonomous motivation, diabetes distress, depression, self-efficacy for diabetes self-care, and neighborhood related stress at baseline (T1) and upon completion of the 6-week intervention at time 2 (T2).

Intervention Week 1. Education and Fitbit set-up/instructions. The women will begin the intervention as soon as five women are enrolled and T1 assessments are completed. The investigators chose the group setting for the education to encourage social interaction and support, which has been associated with DSM in a similar population to ours. The education will consist of two 2-3-hour blocks of interactive diabetes education that will be personalized in response to the cluster members' DM knowledge, health, and self-care history. Education will follow the 2017 National Standards for Diabetes Self-Management and Support. Education sessions will be culturally adapted to reflect needs of AA participants, including feelings of powerlessness, access to care and family roles. Dr. Fritschi (PI) is a certified diabetes educator (CDE) and has worked with low-income, urban diabetes patients since 1994. She will adapt and deliver the education.

Session 1 (2-3 hours): Diabetes self-management education (DSME) will include target glucose ranges, medications, foot care, and dietary and exercise effects on glucose levels.

Session 2 (2-3 hours): At the start of the session, subjects will be given a wrist-worn activity tracker (Fitbit Charge 3 accelerometer) that will be able to assess real-time steps and heart rate. The Fitbit will also be able to track specific activities (e.g., cycling, yoga) that the participant may choose to track. Participants will be taught how to download the Fitbit app into their smart phones and set up personal accounts. The Fitbit Charge 3 was chosen because it has a larger screen and easier app than other devices, and Co-investigator Dr. Ulf Bronas has used the Fitbit extensively in his prior research. Group education will include interactive, hands-on learning about performing foot checks prior to walking; stretching exercises; and creative methods for accumulating steps when the weather or environment doesn't permit walking outside. Participants will individually meet with the exercise physiologist (Dr. Bronas) for a practical educational session using a treadmill-walking bout to determine heart rate goals for moderate and brisk walking. They will be given a written, personalized exercise plan for steps and target heart rate. The group will be coached in setting SMART (specific, measurable, achievable, relevant, and time-bound) goals for the following week. The goals may include Fitbit data, such as goals for step counts, stairs climbed, or minutes of activity.

The Fitbit is a cost-effective wrist-worn activity tracker that is commercially available. Fitbit data provide information on daily level of physical activities and heart rate. Measures include number of steps taken, four levels of activity (sedentary, light, moderate, and moderate-vigorous), distance traveled, and an activity score. Fitbits have been shown to be reliable and valid for step counts and total daily energy expenditure in free-living conditions. The advantages of using a Fitbit tracker are its cost-effectiveness and its ability to measure walking unobtrusively. The investigators are using it as a motivator and an option for individuals to set activity goals. Because patients are more likely to wear the Fitbit continuously, There will be fewer missing data, and activity bouts can be tracked.

Week 2. The women will return to the laboratory for review of their goals and problem-solving sessions with a team member. They will be given a personal-use Freestyle Libre (Abbott Labs, Alameda, CA) Personal CGM (FDA approved). The Libre CGM differs from similar systems in that it is affordable and does not require fingerstick glucose samples for calibration so is not dependent on the user. A small, discrete, water-resistant glucose sensor will be placed on the upper arm by a trained study staff member. The sensor is accurate and stable for up to 14 days. Participants will use a small hand-held "reader" to scan glucose readings whenever they want to, or when prompted. While wearing the CGM, the women will never need to perform a finger stick blood glucose test. Participants will be taught how to use the CGM and how to interpret the graphs that will appear on the reader. Glucose data will be downloaded by our team for analysis of patterns in response to use of the cue cards and Fitbit activity data. Data will also be analyzed for averages of glucose levels by time of day and day; and glucose variability (Standard Deviation). Dr. Fritschi has extensive experience with use of CGM and its data. At the end of the session the women will review their prior goals and may choose to set new goals. The women will work with a member of the team to create a personalized "cue card" that they can carry with them in their pocket or purse. The cue card will be a living document. It will be developed by the study team and the participants and may be revised as necessary.

The cue cards will be approximately the size of a small index card and laminated for durability. One side of the card will have the participants' medications and personal goals. The reverse side of the card will contain a reminder of their target glucose range (80-130 mg/dL), and a list of strategies for activities or eating behaviors they can accomplish within the context of their daily lives. These behavior options will be developed with help from a research team member and other women in their group. At any time during the study, participants may meet with a team member to revise the cue cards. The women will wear their Fitbit and personal CGM continuously for 14-days while using their cue cards. The women will be encouraged to contact the research team for additional problem-solving or questions during this time.

Week 4. The women will return to the laboratory for goal review and problem solving as a group. Data from the Fitbits and CGMs will be downloaded to assess frequency of use, and any device-related problems. Since the CGM sensor is approved for 14-day use only, a new sensor will be attached. At this meeting, the investigators will review and revise the goals based on personal preferences and abilities to meet goals by the women. The goals will be revised as needed. The behaviors may also change. As the women gain experience with the behavior choices, they may decide that the options are too difficult or too easy and thus want to change them. They may have new behavior options they want to try from suggestions made by other women in the group. At the conclusion of the session, new laminated cards will be given to the women.

Weeks 4-6. The women will wear the CGM and Fitbit devices while maintaining their normal routines. Data from each device will be downloaded to assess frequency of use, and any device-related problems.

Week 6. At the end of Week 6, the women will complete T2 assessments and final interviews. The women will be allowed to keep the personal CGM and the Fitbit.

Final Assessments (T2) will include all of the surveys from T1 (excluding health history and eligibility screening). Additionally, the investigators will conduct structured interviews. about the acceptability of the study procedures and suggestions for changes in the intervention for future, larger trials. The interviews will be audio recorded and transcribed by an outside agency. Content analysis will be performed for common themes.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black female
* History of T2DM > 1 year
* Age > 40 years of age
* On non-insulin anti-diabetic therapy or diet-controlled
* Smartphone owner

Exclusion Criteria:

* Women with type 1 diabetes
* Women using insulin
* Any condition that would prohibit the ability to walk for 15-30 minutes or participate in light to moderate physical activity
* Low cognitive function (Mini-cog <3)
* A1c > 10%

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Hours of CGM data | Post-intervention at week 6
  Total number of hours of usable CGM data while worn.
Number of times participants accessed their CGM data | Post-intervention at week 6
  Total number of times the CGM receiver was used to access glucose readings by the participants each day.
Wear time of Fitbit activity monitor | Post-intervention at week 6
  Assessment of wear time will include average hours per day the device was worn.
Interrelationships between real-time interstitial glucose levels (mg/dL) and activity levels (active minutes (correlation coefficients). | Post intervention at week 6
  Correlations between averaged daily glucose levels and average daily active minutes.
Interrelationships between real-time interstitial glucose levels (mg/dL) and activity levels (step counts). | Post intervention at week 6
  Correlations between averaged daily glucose levels and average daily step counts.
Acceptability of intervention: Semi-structured Diabetes Study Acceptability Interview Guide | Post-intervention at week 6
  Semi-structured Diabetes Study Acceptability Interview Guide (developed by investigators). Open-ended questions will address:
  Overall experience; experiences with personalized education; helpfulness of group setting; Difficulty using devices, helpfulness of devices; interference with daily life; and any thoughts or suggestions for changes to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Fritschi, PhD, RN, Principal Investigator — University of Illinois at Chicago, College of Nursing
Locations (1):
- University of Illinois at Chicago, College of Nursing, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No